CLINICAL TRIAL: NCT05823545
Title: Which is Better to Assess Postoperative Complications in Patients Undergoing Laparoscopic Partial Nephrectomy?: Clavien-Dindo Classification Versus Comprehensive Complication Index.
Brief Title: Assessment of Complications in Patients Who Underwent LPN According to the CCI
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Responsible Party: Principal Investigator, Mehmet N. Mercimek, MD, FEBU, Associate professor, MD, FEBU, Samsun Liv Hospital
Other Study IDs: OMU KAEK 26.12.2019/876
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Renal Cancer; Surgery-Complications
Keywords: laparoscopy; partial nephrectomy; complication; CCI; urology
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the strength of the classical Clavien-Dindo classification system (CDC), which is a Likert scale analysis versus the comprehensive complication index (CCI), a new quantitative evaluation system, in patients undergoing laparoscopic partial nephrectomy (LPN).

DETAILED DESCRIPTION:
Prospectively collected data of sixty-two patients undergoing LPN with postoperative complications from November 2009 to August 2020 were evaluated retrospectively. Postoperative complications were classified according to the CDCs and calculated using the CCI calculator (https://www.assessurgery.com) quantitatively. Major complications were determined as ≥ grade 3 complications according to the CDC. The complexity of the renal mass was defined according to the RENAL nephrometry score. The cut-off value for CCI was analyzed by the ROC analysis technique. The significance level was taken as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients with complete data
* patients with consent
* Patients > 18 year-old
* The surgeries performed by the surgeon EO

Exclusion Criteria:

* Missing data
* patients without consent
* patients who underwent open or retroperitoneoscopic laparoscopic partial nephrectomy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A retrospective analysis was carried out on 517 surgical procedures in 503 patients who underwent LPN between November 2009 and August 2020 in a tertiary university hospital. Sixty-two patients with postoperative complications were included in the study.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Postoperative complication | up to 3 months, postoperatively
  Abnormal clinical and laboratory findings that may be seen after surgery and require additional intervention, treatment, or follow-up
Opertaion time | during the surgery (minute)
  From first trocar incision to closure of all incisions
Estimeted blood loss | during the surgery (mL)
  perioperative estimated blood loss
warm ischemia time | during the surgery (minute)
  Its starts when the renal artery and vein are controlled and it ends when reperfusion of the graft kidney starts on the back table

CONTACTS AND LOCATIONS:
Overall Officials: Ender Ozden, Prof., Study Chair — Ondokuz Mayıs University, Faculty of Medicine, Department of Urology; Mehmet N Mercimek, Assoc. Prof., Principal Investigator — Atasam Hospital, Departmen of Urology, Samsun, Turkey
Locations (1):
- Ondokuz Mayıs University, Department of Urology, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loffel LM, Gross T, Schneider MP, Burkhard FC, Thalmann GN, Bosshard P, Wuethrich PY, Furrer MA. Complication reporting with the Bern Comprehensive Complication Index CCI after open radical prostatectomy: A longitudinal long-term single-center study. Urol Oncol. 2020 Mar;38(3):79.e1-79.e8. doi: 10.1016/j.urolonc.2019.09.021. Epub 2019 Dec 31. PMID 31899103
- [Result] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846
- [Result] Kim TH, Suh YS, Huh YJ, Son YG, Park JH, Yang JY, Kong SH, Ahn HS, Lee HJ, Slankamenac K, Clavien PA, Yang HK. The comprehensive complication index (CCI) is a more sensitive complication index than the conventional Clavien-Dindo classification in radical gastric cancer surgery. Gastric Cancer. 2018 Jan;21(1):171-181. doi: 10.1007/s10120-017-0728-3. Epub 2017 Jun 8. PMID 28597328
- See also: Surgical technique — https://pubmed.ncbi.nlm.nih.gov/32967451/